CLINICAL TRIAL: NCT00507143
Title: A Clinical Study for the Evaluation of Genetic Polymorphisms of Drug Transporters and Orphan Nuclear Receptors on the Pharmacokinetics and Treatment Effects of Irinotecan in Patients With Colorectal and Gastric Cancer
Brief Title: Study of Genetic Polymorphisms of Drug Transporters and Orphan Nuclear Receptors on Treatment Effects of Irinotecan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NCCCTS-06-206
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Colorectal Neoplasms; Secondary
Keywords: Colorectal neoplasms; Secondary; irinotecan; Pharmacokinetics; Pharmacodynamics; SLCO1B1; PXR
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: irinotecan

SUMMARY:
From 100 colorectal cancer patients being treated with FOLFIRI regimen or any kind of irinotecan containing regimen, blood samples for irinotecan and its metabolites levels and genotypes related with its metabolism will be collected. The association of their levels and genotypes and treatment effects will be evaluated.

DETAILED DESCRIPTION:
For the genotype-PD association, 50 colorectal cancer patients treated with FOLFIRI will be enrolled and studied. 50 additional colorectal patients treated with any kind of irinotecan containing regimen will be enrolled and including the 50 patients for the genotype-PD association, a total of 100 patients will be evaluated for the genotype-PK association.

Blood samples for PK analysis will be collected from patients with colorectal cancer during 1st treatment cycle of irinotecan and 2nd, 3rd infusion. During the 1st treatment cycle, blood will be drawn 0 h (before irinotecan infusion), 0.75 h, 1.5 h and each at time ranges of 2~8 h, 8~16 h, 24~32h and 48~52 hours after the start of irinotecan infusion over 90 min and additional blood will be collected 48~52 hours after the respective 2nd and 3rd infusion.

For 50 colorectal cancer patient treated with FOLFIRI regimen, responses to the treatment will be assessed every 3 cycles. All assessments will be repeated at the end of trial therapy.

The RECIST criteria for measurable disease will be followed and toxicity will be evaluated according to NCI common toxicity criteria version 3.0.

Time to disease progression will be calculated from the date of study entry to the first objective documentation of progressive disease. Response duration will be measured from the date a patient first fulfills the CR or PR criteria to the first date of objective documentation of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosed unresectable or metastatic colorectal cancer
* Performance status of 0, 1 and 2 on the ECOG criteria
* Disease status must be that of measurable disease as defined by RECIST criteria (For genotype-PD study only) Only non-target lesions are allowed for PK study
* No previous chemotherapy, radiotherapy on the target lesion, immunotherapy; adjuvant chemotherapy with fluoropyrimidines completed at least 6 months ago is allowed (For genotype-PD study only) Previously treated patients are allowed for PK study
* Life expectancy of more than 3 months (For genotype-PD study only)
* Adequate major organ functions
* Compliant patient who can be followed-up adequately
* Informed consent

Exclusion Criteria:

* Active or uncontrolled infection
* Pregnant or breast-feeding women
* Patients with systemic disease, especially cardiovascular disease, who cannot tolerate systemic chemotherapy
* Patients with brain metastasis (For genotype-PD study only)
* Patients treated with radiotherapy within 2 weeks (For genotype-PD study only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-08; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
SLCO1B1 and PXR genotypes and maximal response rate | Before & during treatment
SLCO1B1 and PXR genotypes and pharmacokinetics of SN-38 | Before and 1st cycle

SECONDARY OUTCOMES:
SLCO1B1 and PXR genotypes and response duration, time to progression and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hae Jung, M.D., Principal Investigator
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea